CLINICAL TRIAL: NCT02447003
Title: A Phase II Clinical Trial of Pembrolizumab (MK-3475) as Monotherapy for Metastatic Triple-Negative Breast Cancer (mTNBC) - (KEYNOTE-086)
Brief Title: Study of Pembrolizumab (MK-3475) Monotherapy for Metastatic Triple-Negative Breast Cancer (MK-3475-086/KEYNOTE-086)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-086; 2015-000294-13 (EudraCT Number); 152987 (Registry Identifier: JAPIC)
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Breast Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Pembrolizumab (Experimental): Participants in Cohort A previously received at least one prior systemic treatment for metastatic breast cancer. Participants will be administered pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles (up to ~ 2 years).
  Interventions: Biological: Pembrolizumab
- Cohort B: Pembrolizumab (Experimental): Participants in Cohort B previously received no prior systemic treatment for metastatic breast cancer AND had a programmed cell death-ligand 1 (PD-L1) positive tumor expression. Participants will be administered pembrolizumab 200 mg IV on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles (up to ~ 2 years).
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion of 200 mg.
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
This is a two-part study of pembrolizumab monotherapy in participants with metastatic triple-negative breast cancer (mTNBC). Part 1 of the study will examine the efficacy and safety of pembrolizumab monotherapy as first line or above treatment in participants who have received either no prior systemic treatment or at least one prior systemic treatment for metastatic breast cancer. Part 2 of the study, if done, will expand the investigation of pembrolizumab treatment in a subgroup of participants from Part 1 and will only start after enrollment in Part 1 has been completed. There will be no hypothesis testing in this study.

DETAILED DESCRIPTION:
Qualified participants who complete up to ~2 years of pembrolizumab treatment but progress after discontinuation may be eligible for a second course of pembrolizumab for up to ~1 additional year, at the Investigator's discretion. Per protocol, response or progression during this second course will not count towards efficacy outcome measure and adverse events during this second course will not count towards safety outcome measures.

ELIGIBILITY:
Inclusion Criteria:

For the purposes of this study, neoadjuvant and/or adjuvant chemotherapy regimens do not count as a prior line of therapy.

For second line plus monotherapy (Parts 1 and 2):

* Has received at least one systemic treatment for metastatic breast cancer
* Has documented disease progression on or after the most recent therapy
* Prior treatment must include an anthracycline and a taxane in the neoadjuvant, adjuvant, or metastatic setting

For first line monotherapy (Part 1):

* Has received no prior systemic treatment for metastatic breast cancer
* Has PD-L1-positive mTNBC.

For second line plus monotherapy (Part 2):

- Has PD-L1 strong positive mTNBC

For all parts:

* Has mTNBC confirmed by a central laboratory
* For biomarker analysis, adequate newly obtained core or excisional biopsy of a not-previously-irradiated metastatic tumor lesion (mandatory)
* Has measurable metastatic disease
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Female participants of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study treatment
* Male participants should agree to use an adequate method of contraception starting with the first dose of study treatment through 120 days after the last dose of study treatment
* Has adequate organ function

Exclusion Criteria:

* Is currently participating and receiving study treatment, or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to study Day 1
* Has received prior anti-cancer monoclonal antibody (mAb) therapy for direct anti-neoplastic treatment within 4 weeks prior to study Day 1
* Has received prior chemotherapy, targeted small molecule therapy, or radiation therapy within at least 2 weeks prior to study Day 1
* Has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered within at least 2 weeks prior to study Day 1
* Has an active autoimmune disease requiring systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Has known additional malignancy that progressed or required active treatment within the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer
* Has radiographically-detectable central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis or a history of interstitial lung disease
* Has an active infection requiring systemic therapy
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has received prior therapy with an anti-programmed cell death protein-1 (anti-PD-1), anti-PD-L1, anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein-4 [CTLA-4], OX-40, CD137) or has participated in Merck MK-3475 (pembrolizumab) study
* Has a known history of human immunodeficiency virus (HIV)
* Has known active Hepatitis B or C
* Has received a live vaccine within 30 days of planned start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Loi S, Salgado R, Schmid P, Cortes J, Cescon DW, Winer EP, Toppmeyer DL, Rugo HS, De Laurentiis M, Nanda R, Iwata H, Awada A, Tan AR, Sun Y, Karantza V, Wang A, Huang L, Saadatpour A, Cristescu R, Yearley J, Lunceford J, Jelinic P, Adams S. Association Between Biomarkers and Clinical Outcomes of Pembrolizumab Monotherapy in Patients With Metastatic Triple-Negative Breast Cancer: KEYNOTE-086 Exploratory Analysis. JCO Precis Oncol. 2023 Apr;7:e2200317. doi: 10.1200/PO.22.00317. PMID 37099733
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- [Derived] Adams S, Schmid P, Rugo HS, Winer EP, Loirat D, Awada A, Cescon DW, Iwata H, Campone M, Nanda R, Hui R, Curigliano G, Toppmeyer D, O'Shaughnessy J, Loi S, Paluch-Shimon S, Tan AR, Card D, Zhao J, Karantza V, Cortes J. Pembrolizumab monotherapy for previously treated metastatic triple-negative breast cancer: cohort A of the phase II KEYNOTE-086 study. Ann Oncol. 2019 Mar 1;30(3):397-404. doi: 10.1093/annonc/mdy517. PMID 30475950
- [Derived] Adams S, Loi S, Toppmeyer D, Cescon DW, De Laurentiis M, Nanda R, Winer EP, Mukai H, Tamura K, Armstrong A, Liu MC, Iwata H, Ryvo L, Wimberger P, Rugo HS, Tan AR, Jia L, Ding Y, Karantza V, Schmid P. Pembrolizumab monotherapy for previously untreated, PD-L1-positive, metastatic triple-negative breast cancer: cohort B of the phase II KEYNOTE-086 study. Ann Oncol. 2019 Mar 1;30(3):405-411. doi: 10.1093/annonc/mdy518. PMID 30475947
- [Derived] Nanda R, Chow LQ, Dees EC, Berger R, Gupta S, Geva R, Pusztai L, Pathiraja K, Aktan G, Cheng JD, Karantza V, Buisseret L. Pembrolizumab in Patients With Advanced Triple-Negative Breast Cancer: Phase Ib KEYNOTE-012 Study. J Clin Oncol. 2016 Jul 20;34(21):2460-7. doi: 10.1200/JCO.2015.64.8931. Epub 2016 May 2. PMID 27138582
- See also: Merck Oncology Clinical Trial Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, response or progression during the second pembrolizumab course was not counted towards efficacy outcome measures, and adverse events during the second pembrolizumab course were not counted towards safety outcome measures.
  Based on protocol-specified inclusion criteria and outcome analyses requirements, Part 2 was not conducted.
Groups:
- Cohort A: Pembrolizumab: Participants in Cohort A previously received at least one prior systemic treatment for metastatic breast cancer. Participants were administered pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles (up to ~2 years). Qualified participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 each 3-week cycle (Q3W), for up to 17 cycles (up to ~1 year).
- Cohort B: Pembrolizumab: Participants in Cohort B previously received no prior systemic treatment for metastatic breast cancer AND had a programmed cell death-ligand 1 (PD-L1) positive tumor expression. Participants were administered pembrolizumab 200 mg IV on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles (up to ~2 years). Qualified participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 of each 3-week cycle (Q3W), for up to 17 cycles (up to ~1 year).
Period: Overall Study
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Started | 170 | 84
Completed | 0 | 0
Not Completed | 170 | 84
Not completed — Other | 0 | 4
Not completed — Site discontinued | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Sponsor Decision | 6 | 11
Not completed — Progressive Disease | 1 | 0
Not completed — Lost to Follow-up | 5 | 0
Not completed — Death | 154 | 63

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab | Total
Number analyzed (Participants) | 170 | 84 | 254
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (12.8) | 54.2 (14.1) | 54.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 84 | 254
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 146 | 74 | 220
  Unknown or Not Reported | 14 | 4 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 24 | 15 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 14 | 26
  White | 129 | 53 | 182
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Central Imaging Vendor (CIV) in All Cohort A Participants
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in sum of diameters [SOD] of target lesions) per RECIST 1.1 by CIV. ORR was estimated by Agresti-Coull (A-C) method. The percentage of participants who had CR or PR is reported here as the protocol-specified ORR, for the first pembrolizumab course, assessed from enrolment/treatment initiation and analyzed by Cohort, for all participants in Cohort A. Per protocol final ORR analysis in all Cohort A participants was done at the time of final statistical efficacy analysis, with a 10-November (Nov)-2017 cutoff. Per protocol ORR per RECIST 1.1 by CIV in all Cohort A participants was planned and conducted as a pre-specified primary outcome analysis. Per protocol ORR per RECIST 1.1 by CIV in all Cohort B participants was analyzed separately as a pre-specified secondary outcome analysis and reported later in the record.
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol ORR, for the first pembrolizumab course, was analyzed by Cohort in all participants in Cohort A who got ≥1 dose of study drug. Per protocol ORR per RECIST 1.1 by CIV was analyzed separately in all Cohort B participants as a pre-specified secondary outcome analysis and is not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort A: Pembrolizumab: Participants in Cohort A previously received at least one prior systemic treatment for metastatic breast cancer. Participants were administered pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles (up to ~2 years).
- Cohort B: Pembrolizumab: Participants in Cohort B previously received no prior systemic treatment for metastatic breast cancer AND had a programmed cell death-ligand 1 (PD-L1) positive tumor expression. Participants were administered pembrolizumab 200 mg IV on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles (up to ~2 years).
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 170 | 0
Percentage of participants | 5.3 [2.7 to 9.9] |

2. Primary Outcome: ORR Per RECIST 1.1 by CIV in Subgroup of Cohort A Participants With Programmed Cell Death- Ligand 1 (PD-L1) Positive Tumor Expression
Description: ORR was defined as the percentage of participants who had a CR (disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 by CIV. ORR was estimated by A-C method. The percentage of participants who had CR or PR is reported here as the protocol-specified ORR, for the first pembrolizumab course, assessed from enrolment/treatment initiation and analyzed by Cohort for the subgroup of Cohort A participants with tumor immunohistochemistry (IHC) defined-PD-L1 positive expression (PD-L1+). Per protocol final ORR analysis in the Cohort A PD-L1+ subgroup was done at the time of final statistical efficacy analysis with a 10-Nov-2017 cutoff. Per protocol all Cohort B participants were PD-L1+ and ORR per RECIST 1.1 by CIV in all Cohort B participants was analyzed separately as a pre-specified secondary outcome analysis and reported later in the record.
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol ORR for the first pembrolizumab course, was analyzed by Cohort in the subgroup of Cohort A participants who were PD-L1+ and got ≥1 dose of study drug. Per protocol all Cohort B participants were PD-L1+; per protocol ORR per RECIST 1.1 by CIV was analyzed separately in all Cohort B participants as a pre-specified secondary outcome analysis and is not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 105 | 0
Percentage of participants | 5.7 [2.4 to 12.2] |

3. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that is temporally associated with the use of the Sponsor's product is also an AE. Per protocol the number of participants who experienced at least one AE, for the first pembrolizumab course, was assessed from enrollment/treatment initiation of a participant and analyzed by Cohort and is reported here for all participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Time Frame: Up to ~31 months
Population: Per protocol participants who experienced AEs, for the first pembrolizumab course, were analyzed by Cohort in all participants in Cohort A and Cohort B who got ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 170 | 84
Participants | 161 | 83

4. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that is temporally associated with the use of the Sponsor's product is also an AE. Per protocol the number of participants who discontinued study drug due to an AE, in the first pembrolizumab course, was assessed from enrolment/treatment initiation of a participant and analyzed by Cohort and is reported here for all participants in Cohort A and Cohort B who received ≥1 dose of study drug.
Time Frame: Up to ~31 months
Population: Per protocol participants who discontinued study drug due to an AE, for the first pembrolizumab course, were analyzed by Cohort in all participants in Cohort A and Cohort B who got ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 170 | 84
Participants | 8 | 3

5. Secondary Outcome: ORR Per RECIST 1.1 by CIV in All Cohort B Participants
Description: ORR was defined as the percentage of participants who had a CR (disappearance of all target lesions) or a PR (≥30% decrease in SOD of target lesions) per RECIST 1.1 by CIV. ORR was estimated by A-C method. The percentage of participants who had CR or PR is reported here as the protocol-specified ORR, for the first pembrolizumab course, assessed from enrolment/treatment initiation and analyzed by Cohort for all participants in Cohort B. Per protocol final ORR analysis in all Cohort B participants was done at the time of final statistical efficacy analysis, with a 10-Nov-2017 cutoff. Per protocol ORR per RECIST 1.1 by CIV in all Cohort B participants was planned and conducted as a pre-specified secondary outcome analysis. Per protocol ORR per RECIST 1.1 by CIV in all Cohort A participants was analyzed separately as a pre-specified primary outcome analysis and reported earlier in the record.
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol ORR, for the first pembrolizumab course, was analyzed by Cohort in all participants in Cohort B who got ≥1 dose of study drug. Per protocol ORR per RECIST 1.1 by CIV was analyzed separately in all Cohort A participants as a pre-specified primary outcome analysis and is not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 0 | 84
Percentage of participants |  | 21.4 [13.9 to 31.4]

6. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 by CIV in All Cohort A and Cohort B Participants
Description: For participants who had CR (disappearance of all target lesions) or PR (≥30% target lesion SOD decrease) per RECIST 1.1 by CIV, DOR was defined as time from first documented CR or PR until progressive disease (PD: ≥20% target lesion SOD increase, ≥5 mm absolute SOD increase; PD is also ≥1 new lesion appearance) or death. DOR for those who didn't progress/die at time of analysis was censored at last tumor assessment. Per protocol DOR for the first pembrolizumab course, assessed from enrolment/treatment initiation, estimated by Kaplan-Meier (KM) method and analyzed by cohort is reported here for all participants in Cohort A and Cohort B who had CR or PR per RECIST 1.1 by CIV. Per protocol final DOR analysis in all Cohort A and Cohort B participants was done at the time of final statistical efficacy analysis with a 10-Nov-2017 cutoff.
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol DOR, for the first pembrolizumab course, was analyzed by Cohort in all participants in Cohort A and Cohort B who had CR or PR per RECIST 1.1 by CIV and got ≥1 dose of study drug.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 9 | 18
Months | NA [NA to NA] — Median and range lower and upper limit not reached (no progressive disease by the time of last disease assessment) | 10.4 [4.2 to NA] — Range upper limit not reached (no progressive disease by the time of last disease assessment)

7. Secondary Outcome: DOR Per RECIST 1.1 by CIV in Subgroup of Cohort A Participants With PD-L1 Positive Tumor Expression
Description: For participants who had CR (disappearance of all target lesions) or PR (≥30% target lesion SOD decrease) per RECIST 1.1 by CIV, DOR was defined as time from first documented CR or PR until PD (≥20% target lesion SOD increase, ≥5 mm absolute SOD increase; PD is also ≥1 new lesion appearance) or death. DOR for those who didn't progress/die at time of analysis was censored at last tumor assessment. Per protocol DOR for first pembrolizumab course, assessed from enrolment/treatment initiation, estimated by KM method and analyzed by Cohort is reported here for subgroup of Cohort A participants with tumor IHC defined-PD-L1 positive expression (PD-L1+) and CR/PR per RECIST 1.1 by CIV. Per protocol final DOR analysis in Cohort A PD-L1+ subgroup was done at time of final statistical efficacy analysis with a 10-Nov-2017 cutoff. Per protocol all Cohort B participants were PD-L1+ and DOR per RECIST 1.1 by CIV in all Cohort B participants was analyzed separately and reported earlier in the record
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol DOR, for the first pembrolizumab course, was analyzed by Cohort in the subgroup of Cohort A participants who were PD-L1+, had CR or PR per RECIST 1.1 by CIV and got ≥1 dose of study drug. Per protocol all Cohort B participants were PD-L1+; per protocol DOR per RECIST 1.1 by CIV was analyzed separately in all Cohort B participants and is not included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 6 | 0
Months | NA [6.3 to NA] — Median and range upper limit not reached (no progressive disease by the time of last disease assessment) |

8. Secondary Outcome: Disease Control Rate (DCR) Per RECIST 1.1 by CIV in All Cohort A and Cohort B Participants
Description: DCR was defined as the percentage of participants in the analysis population who have CR (disappearance of all target lesions) or PR (≥30% target lesion SOD decrease) or SD (not sufficient shrinkage for PR or sufficient increase for PD [≥20% target lesion SOD increase, ≥5 mm absolute SOD increase; PD is also ≥1 new lesion appearance]) for ≥24 weeks per RECIST 1.1 by CIV. Per protocol percentage of participants who had CR, PR or SD per RECIST 1.1 by CIV is reported here as DCR, for the first pembrolizumab course, assessed from enrolment/treatment initiation, estimated by A-C method and analyzed by Cohort, for all participants in Cohort A and Cohort B. Per protocol final DCR analysis in all Cohort A and Cohort B participants was done at the time of final statistical efficacy analysis, with a 10-Nov-2017 cutoff.
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol DCR, for the first pembrolizumab course, was analyzed by Cohort in all participants in Cohort A and Cohort B who got ≥1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 170 | 84
Percentage of participants | 7.6 [4.4 to 12.7] | 23.8 [15.9 to 34.0]

9. Secondary Outcome: DCR Per RECIST 1.1 by CIV in Subgroup of Cohort A Participants With PD-L1 Positive Tumor Expression
Description: DCR was defined as the percentage of participants who have CR (disappearance of all target lesions) or PR (≥30% target lesion SOD decrease) or SD (not sufficient shrinkage for PR or sufficient increase for PD [≥20% target lesion SOD increase, ≥5 mm absolute SOD increase; PD is also ≥1 new lesion appearance]) for ≥24 weeks per RECIST 1.1 by CIV. Per protocol percentage of participants who had CR, PR or SD per RECIST 1.1 by CIV is reported here as DCR for the first pembrolizumab course, assessed from enrolment/treatment initiation, estimated by A-C method and analyzed by Cohort for subgroup of Cohort A participants with tumor IHC defined-PD-L1 positive expression (PD-L1+). Per protocol final DCR analysis in Cohort A PD-L1+ subgroup was done at the time of final statistical efficacy analysis with a 10-Nov-2017 cutoff. Per protocol all Cohort B participants were PD-L1+ and DCR per RECIST 1.1 by CIV in all Cohort B participants was analyzed separately and reported earlier in the record.
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol DCR, for the first pembrolizumab course, was analyzed by Cohort in the subgroup of Cohort A participants who were PD-L1+ and got ≥1 dose of study drug. Per protocol all Cohort B participants were PD-L1+; per protocol DCR per RECIST 1.1 by CIV was analyzed separately in all Cohort B participants and is not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 105 | 0
Percentage of participants | 9.5 [5.1 to 16.8] |

10. Secondary Outcome: Progression Free Survival (PFS) Per RECIST 1.1 by CIV in All Cohort A and Cohort B Participants
Description: PFS was defined as the time from first dose of study drug to the first documented PD per RECIST 1.1 by CIV, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. PFS was estimated by KM method. Per protocol PFS, for the first pembrolizumab course, assessed from enrolment/treatment initiation and analyzed by Cohort is reported here for all participants in Cohort A and Cohort B. Per protocol final PFS analysis in all Cohort A and Cohort B participants was done at the time of final statistical efficacy analysis with a 10-Nov-2017 cutoff.
Time Frame: Up to ~28 months (through pre-specified final statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol PFS, for the first pembrolizumab course, was analyzed by Cohort in all participants in Cohort A and Cohort B who got ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 170 | 84
Months | 2.0 [1.9 to 2.0] | 2.1 [2.0 to 2.2]

11. Secondary Outcome: PFS Per RECIST 1.1 by CIV in Subgroup of Cohort A Participants With PD-L1 Positive Tumor Expression
Description: PFS was defined as the time from first dose of study drug to the first documented PD per RECIST 1.1 by CIV, or death due to any cause, whichever occurred first. Per RECIST 1.1 PD was defined as ≥20% increase in SOD of target lesions and absolute SOD increase of ≥5 mm. Appearance of ≥1 new lesion is also PD. PFS was estimated by KM method. Per protocol PFS, for the first pembrolizumab course, assessed from enrolment/treatment initiation and analyzed by Cohort is reported here for the subgroup of Cohort A participants with tumor IHC defined-PD-L1 positive expression (PD-L1+). Per protocol final PFS analysis in the Cohort A PD-L1+ subgroup was done at the time of final statistical efficacy analysis with a 10-Nov-2017 cutoff. Per protocol all Cohort B participants were PD-L1+ and PFS per RECIST 1.1 by CIV in all Cohort B participants was analyzed separately and reported earlier in the record.
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol PFS, for the first pembrolizumab course, was analyzed by Cohort in the subgroup of Cohort A participants who were PD-L1+ and got ≥1 dose of study drug. Per protocol all Cohort B participants were PD-L1+; per protocol PFS per RECIST 1.1 by CIV was analyzed separately in all Cohort B participants and is not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 105 | 0
Months | 2.0 [1.9 to 2.1] |

12. Secondary Outcome: Overall Survival (OS) in All Cohort A and Cohort B Participants
Description: OS was defined as the time from the first dose of study drug to death due to any cause. OS was estimated by KM method. Per protocol OS, for the first pembrolizumab course, assessed from enrolment/treatment initiation and analyzed by Cohort is reported here for all participants in Cohort A and Cohort B. Per protocol final OS analysis in all Cohort A and Cohort B participants was done at the time of final statistical efficacy analysis with a 10-Nov-2017 cutoff.
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol OS, for the first pembrolizumab course, was analyzed by Cohort in all participants in Cohort A and Cohort B who got ≥1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 170 | 84
Months | 9.0 [7.6 to 11.2] | 18.0 [12.9 to 23.0]

13. Secondary Outcome: OS in Subgroup of Cohort A Participants With PD-L1 Positive Tumor Expression
Description: OS was defined as the time from the first dose of study drug to death due to any cause. OS was estimated by KM method. Per protocol OS, for the first pembrolizumab course, assessed from enrolment/treatment initiation and analyzed by Cohort, is reported here for the subgroup of Cohort A participants with tumor IHC defined-PD-L1 positive expression (PD-L1+). Per protocol final OS analysis in the Cohort A PD-L1+ subgroup was done at the time of final statistical efficacy analysis with a 10-Nov-2017 cutoff. Per protocol all Cohort B participants were PD-L1+ and OS in all Cohort B participants was analyzed separately and reported earlier in the record.
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol OS for the first pembrolizumab course, was analyzed by Cohort in the subgroup of Cohort A participants who were PD-L1+ and got ≥1 dose of study drug. Per protocol all Cohort B participants were PD-L1+; per protocol OS was analyzed separately in all Cohort B participants and is not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 105 | 0
Months | 8.8 [7.1 to 11.2] |

14. Secondary Outcome: Odds Ratio of Association Between PD-L1 Tumor Expression and Objective Response (OR) Per RECIST 1.1 by CIV in Cohort A Participants
Description: OR comprises CR (disappearance of all target lesions) or PR (≥30% target lesion SOD decrease) per RECIST 1.1 by CIV. PD-L1 expression is assessed by IHC-defined combined positive score (CPS). Association between (b/w) PD-L1 CPS and OR was assessed by odds ratio using a logistic regression model and was calculated as ratio of odds of OR per unit CPS increase in a single arm (odds ratio=1: no association; odds ratio<1: negative association [increase in CPS lowers odds of OR]; odds ratio >1: positive association [increase in CPS raises odds of OR]). Per protocol odds ratio, for the first pembrolizumab course, assessed from enrolment/treatment initiation and analyzed by Cohort is reported here in a single arm of Cohort A participants with PD-L1 CPS available. Per protocol odds ratio was analyzed at the time of final statistical efficacy analysis with a 10-Nov-2017 cutoff. Per protocol odds ratio of association b/w PD-L1 expression and OR was not planned or done in Cohort B participants.
Time Frame: Up to ~28 months (through pre-specified statistical analysis cut-off date of 10-Nov-2017)
Population: Per protocol odds ratio, for the first pembrolizumab course, was analyzed by Cohort in all participants in Cohort A who got ≥1 dose of study drug and had CPS for PD-L1 available. Per protocol odds ratio of association b/w PD-L1 expression and OR was not planned or conducted in cohort B participants.
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Cohort A: Pembrolizumab | Cohort B: Pembrolizumab
Number analyzed (Participants) | 169 | 0
Odds Ratio | 1.017 [0.991 to 1.043] |

ADVERSE EVENTS:
Time Frame: Safety: Up to ~31 months for pembrolizumab first course and up to additional ~15 months for pembrolizumab second course (AEs were collected through 90 days post treatment for SAEs and 30 days post treatment for NSAEs); All-cause mortality (ACM): Up to ~54 months for pembrolizumab first and second course
Description: Safety and ACM were analyzed by Cohort (A and B) and by Course of pembrolizumab (first and second course) in all participants who got ≥1 dose of study drug, and were assessed from a participant's enrolment/treatment initiation. Per protocol disease progression of cancer was not considered an AE unless considered related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Cohort A: Pembrolizumab First Course: Participants in Cohort A previously received at least one prior systemic treatment for metastatic breast cancer. Participants were administered pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles (up to ~2 years).
- Cohort A: Pembrolizumab Second Course: Qualified Cohort A participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 each 3-week cycle (Q3W) for up to 17 cycles (up to ~1 year).
- Cohort B: Pembrolizumab First Course: Participants in Cohort B previously received no prior systemic treatment for metastatic breast cancer AND had a programmed cell death-ligand 1 (PD-L1) positive tumor expression. Participants were administered pembrolizumab 200 mg IV on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles (up to ~2 years).
- Cohort B: Pembrolizumab Second Course: Qualified Cohort B participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 of each 3-week cycle (Q3W) for up to 17 cycles (up to ~1 year).
Arm/Group | Cohort A: Pembrolizumab First Course | Cohort A: Pembrolizumab Second Course | Cohort B: Pembrolizumab First Course | Cohort B: Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 154/170 | 0/1 | 63/84 | 0/4
Serious Adverse Events (participants affected / at risk) | 46/170 | 0/1 | 19/84 | 2/4
Other Adverse Events (participants affected / at risk) | 147/170 | 1/1 | 79/84 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Pembrolizumab First Course (N=170) | Cohort A: Pembrolizumab Second Course (N=1) | Cohort B: Pembrolizumab First Course (N=84) | Cohort B: Pembrolizumab Second Course (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (7) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device failure (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0) | 3 (5) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Pembrolizumab First Course (N=170) | Cohort A: Pembrolizumab Second Course (N=1) | Cohort B: Pembrolizumab First Course (N=84) | Cohort B: Pembrolizumab Second Course (N=4)
Anaemia (Blood and lymphatic system disorders) | 18 (22) | 0 (0) | 10 (12) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 9 (9) | 0 (0) | 4 (5) | 0 (0)
Hypothyroidism (Endocrine disorders) | 19 (20) | 0 (0) | 9 (10) | 1 (1)
Vision blurred (Eye disorders) | 3 (3) | 0 (0) | 5 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 0 (0) | 9 (14) | 1 (1)
Constipation (Gastrointestinal disorders) | 33 (36) | 0 (0) | 9 (11) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 22 (32) | 0 (0) | 16 (24) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 11 (11) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 34 (41) | 0 (0) | 23 (29) | 0 (0)
Vomiting (Gastrointestinal disorders) | 19 (24) | 0 (0) | 11 (21) | 0 (0)
Asthenia (General disorders) | 19 (20) | 0 (0) | 8 (9) | 1 (1)
Chest pain (General disorders) | 11 (13) | 0 (0) | 6 (7) | 0 (0)
Fatigue (General disorders) | 49 (59) | 0 (0) | 30 (40) | 1 (1)
Oedema peripheral (General disorders) | 15 (18) | 0 (0) | 7 (8) | 0 (0)
Pain (General disorders) | 5 (5) | 0 (0) | 5 (5) | 0 (0)
Pyrexia (General disorders) | 19 (25) | 0 (0) | 10 (12) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (8) | 0 (0) | 6 (6) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0) | 7 (7) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (7) | 0 (0) | 6 (7) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 12 (14) | 0 (0) | 8 (9) | 1 (1)
Weight decreased (Investigations) | 10 (10) | 0 (0) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 28 (30) | 0 (0) | 12 (14) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (38) | 0 (0) | 15 (20) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 0 (0) | 16 (19) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 0 (0) | 4 (4) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 0 (0) | 6 (7) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (14) | 0 (0) | 9 (10) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (18) | 1 (1) | 7 (9) | 0 (0)
Dizziness (Nervous system disorders) | 11 (11) | 0 (0) | 10 (11) | 0 (0)
Headache (Nervous system disorders) | 13 (16) | 0 (0) | 16 (18) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (4) | 0 (0) | 9 (11) | 0 (0)
Anxiety (Psychiatric disorders) | 11 (11) | 0 (0) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 8 (8) | 0 (0) | 5 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 0 (0) | 7 (7) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 39 (45) | 0 (0) | 20 (22) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 0 (0) | 17 (21) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 0 (0) | 3 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (21) | 0 (0) | 8 (10) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 12 (14) | 0 (0) | 14 (23) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 5 (8) | 0 (0)
Hot flush (Vascular disorders) | 8 (8) | 0 (0) | 6 (6) | 0 (0)
Lymphoedema (Vascular disorders) | 9 (10) | 0 (0) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 2 (2) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 1 (3) | 1 (1)
Weight increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT02447003/Prot_SAP_000.pdf